CLINICAL TRIAL: NCT00295945
Title: Outcomes of Perioperative Epidural Analgesia in Gynecologic Oncology Patients: A Parallel Prospective Cohort and Randomized Clinical Study
Brief Title: Epidural Analgesia or Patient-Controlled Analgesia in Treating Patients Who Have Undergone Surgery for Gynecologic Cancer
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000459963; UCSF-03423 (Other: UCSF CHR); UCSF-H10588-24197-02 (Other: UCSF CHR)
Record Dates: First submitted 2006-02-23; First posted 2006-02-24 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Pain; Perioperative/Postoperative Complications; Sarcoma
Keywords: pain; perioperative/postoperative complications; stage III cervical cancer; recurrent cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IA cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; recurrent endometrial carcinoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; ovarian sarcoma; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; ovarian stromal cancer; recurrent fallopian tube cancer; stage IA fallopian tube cancer; stage IB fallopian tube cancer; stage IC fallopian tube cancer; stage IIA fallopian tube cancer; stage IIB fallopian tube cancer; stage IIC fallopian tube cancer; stage IIIA fallopian tube cancer; stage IIIB fallopian tube cancer; stage IIIC fallopian tube cancer; stage IV fallopian tube cancer; stage IA ovarian epithelial cancer; stage IB ovarian epithelial cancer; stage IC ovarian epithelial cancer; stage IIA ovarian epithelial cancer; stage IIB ovarian epithelial cancer; stage IIC ovarian epithelial cancer; stage IIIA ovarian epithelial cancer; stage IIIB ovarian epithelial cancer; stage IIIC ovarian epithelial cancer; stage IA ovarian germ cell tumor; stage IB ovarian germ cell tumor; stage IC ovarian germ cell tumor; stage IIA ovarian germ cell tumor; stage IIB ovarian germ cell tumor; stage IIC ovarian germ cell tumor; stage IIIA ovarian germ cell tumor; stage IIIB ovarian germ cell tumor; stage IIIC ovarian germ cell tumor
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Pain; Postoperative Complications; Sarcoma; Carcinoma, Ovarian Epithelial | interventions — Fentanyl; Hydromorphone; Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- PCA: Patient-controlled intravenous analgesia
  Interventions: Drug: hydromorphone hydrochloride
- PCEA: Perioperative patient-controlled epidural analgesia
  Interventions: Drug: fentanyl citrate; Drug: ropivacaine hydrochloride

INTERVENTIONS:
Drug: fentanyl citrate
  Groups: PCEA
Drug: hydromorphone hydrochloride
  Groups: PCA
Drug: ropivacaine hydrochloride
  Groups: PCEA

SUMMARY:
RATIONALE: Giving pain medication into the space between the wall of the spinal canal and the covering of the spinal cord or giving it into a vein may help lessen pain caused by cancer surgery. It is not yet known whether epidural analgesia is more effective than patient-controlled analgesia in controlling pain in patients who have undergone surgery for gynecologic cancer.

PURPOSE: This randomized clinical trial is studying epidural analgesia to see how well it works compared to patient-controlled analgesia in treating patients who have undergone surgery for gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the gradual weaning of an epidural opioid can shorten the duration of postoperative ileus, without worsening pain control, in patients who have undergone surgery for gynecologic cancer.
* Compare postoperative pain management in patients treated with perioperative epidural analgesia vs patient controlled analgesia.
* Compare time to ambulation, return of bowel function, and readiness for hospital discharge in patients treated with these pain management interventions.
* Compare the incidence of perioperative complications (e.g., bleeding, hypotension, thromboembolic events, pneumonia, wound infection, myocardial infection, or death) in patients treated with these pain management interventions.

OUTLINE: This is a partially randomized, double-blind, parallel-group study. Patients choose between epidural analgesia or patient controlled analgesia (PCA) for perioperative pain management. Patients for whom an epidural is contraindicated receive a PCA. Patients are assigned to 1 of 2 treatment groups. Patients in group 1 are stratified according to bowel resection surgery (yes vs no) and prior abdominal surgery (yes vs no).

* Group 1 (epidural): Patients undergo placement of a thoracic epidural catheter followed by abdominal/pelvic surgery. Patients then begin an epidural infusion of ropivacaine hydrochloride and fentanyl immediately after surgery (postoperative day 0). Patients may also be supplemented with a patient controlled demand dose. The day after surgery (postoperative day 1), patients are randomized (as long as there is adequate pain control) to 1 of 2 epidural management arms.

  * Arm I: Patients continue to receive the epidural infusion until they can be weaned to oral pain medication.
  * Arm II: Patients undergo daily weaning of the fentanyl concentration of the epidural infusion.
* Group 2 (PCA): Patients begin PCA immediately after undergoing abdominal/pelvic surgery (postoperative day 0). Patients receive a demand schedule of hydromorphone IV until they can be weaned to oral pain medication.

In both groups, the Gynecologic Oncology pain service may make adjustments to the epidural infusion or PCA for optimal pain management until the patient can be weaned to oral pain medication.

PROJECTED ACCRUAL: A total of 224 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a gynecologic malignancy
* Scheduled to undergo open abdominal/pelvic surgery (i.e., laparotomy) on the gynecologic oncology service at the University of California San Francisco Medical Center
* No failed epidural catheters (for patients choosing epidural analgesia)
* No lumbar epidurals (for patients choosing epidural analgesia)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: DISEASE CHARACTERISTICS:
  * Diagnosis of a gynecologic malignancy
  * Scheduled to undergo open abdominal/pelvic surgery (i.e., laparotomy) on the gynecologic oncology service at the University of California San Francisco Medical Center
  * No failed epidural catheters (for patients choosing epidural analgesia)
  * No lumbar epidurals (for patients choosing epidural analgesia)
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Time to return to bowel function at discharge | Days

SECONDARY OUTCOMES:
Pain score daily | Days

CONTACTS AND LOCATIONS:
Overall Officials: Lee-may Chen, MD, Study Chair — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States